CLINICAL TRIAL: NCT01825473
Title: Study of Erythromycin in GER-Associated Apnea of the Newborn
Acronym: SEGAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Faranek Davalian, MD, Neonatology Fellow, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16220
Record Dates: First submitted 2013-03-20; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Gastroesophageal Reflux; Apnea; Bradycardia
Keywords: neonate; apnea; preterm; reflux; gastroesophageal reflux; impedance; erythromycin; desaturation; bradycardia; hypoxia
MeSH Terms: conditions — Gastroesophageal Reflux; Apnea; Bradycardia; Premature Birth; Hypoxia | interventions — Erythromycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erythromycin (Experimental): 50 mg/kg/day divided every 6 hours oral for 7 days
  Interventions: Drug: Erythromycin; Device: Multi-channel intra-luminal impedance (MII) pH monitoring
- Placebo (Placebo Comparator): Dextrose 5 Water (D5W) equal amount as experimental every 6 hours oral for 7 days
  Interventions: Device: Multi-channel intra-luminal impedance (MII) pH monitoring; Drug: Placebo (D5W)

INTERVENTIONS:
Drug: Erythromycin
  Arms: Erythromycin
Device: Multi-channel intra-luminal impedance (MII) pH monitoring
  Other Names: Sandhill 6.5 French, product# ZINBS45E
Drug: Placebo (D5W)
  Arms: Placebo

SUMMARY:
To evaluate the relationship of reflux and apnea and to determine whether the administration of erythromycin improves the incidence of GER and GER-associated apnea, bradycardic and/or desaturation events in a prospective randomized controlled trial.

DETAILED DESCRIPTION:
A randomized placebo-controlled trial to determine whether erythromycin, a drug known to enhance gut motility, will improve the incidence of GER and GER-associated apnea, bradycardiac and/or hypoxic events. The investigators have two aims: 1) to examine the relationship between GER and apnea, bradycardia, and/or desaturation (ABD) events by simultaneously employing a unique computer algorithm developed at the University of Virginia to measure ABD events and an Multi-channel Intra-luminal Impedance (MII) pH monitoring to measure GER episodes. 2) In a randomized placebo-controlled trial, the investigators will study whether erythromycin decreases GER and GER-associated apnea, bradycardia and/or hypoxia in premature infants.

ELIGIBILITY:
Inclusion Criteria:Infants admitted to neonatal intensive care unit who are <37 weeks at birth and >14 days of age, non-intubated, on full feeds for 3 days with one of the following:

* Any apnea, bradycardia, or desaturation (ABD) event, or
* Documented symptoms of reflux

Exclusion Criteria:

* major central nervous system, gastrointestinal, or complex cardiac anomalies

Min Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Reflux Impedance events (both acidic and non-acidic) as recorded by Multichannel Intraluminal (MII) pH Impedance | during day 6 to 7 of study treatment

SECONDARY OUTCOMES:
ABD events per Physiologic Monitoring Database | during the entire 7 days of treatment
  Number of apnea, bradycardia, and/or desaturation events (ABD) per computer algorithm developed at University of Virginia
ABD events recorded by nursing | during the entire 7 days of treatment
  Number of apnea, bradycardia, and/or desaturations (ABD) recorded by bedside nurse

CONTACTS AND LOCATIONS:
Overall Officials: Fara Davalian, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Children's Hospital, Charlottesville, Virginia, United States